CLINICAL TRIAL: NCT01942330
Title: Prospective Evaluation of a Laparoscopic-Assisted Transvaginal Approach for Colonic Resection
Brief Title: Pain and Infection After Transvaginal Colectomy
Acronym: TVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jaime Sanchez (Other)
Responsible Party: Sponsor-Investigator, Jaime Sanchez, Assistant Professor of Surgery, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006972
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Colonic Resection Procedures
MeSH Terms: interventions — Natural Orifice Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Laparoscopic-Assisted Colectomy (No Intervention)
- Transvaginal Laparoscopic-Assisted Colectomy (Experimental): Laparoscopic-Assisted Natural Orifice Surgery
  Interventions: Procedure: Laparoscopic-Assisted Natural Orifice Surgery

INTERVENTIONS:
Procedure: Laparoscopic-Assisted Natural Orifice Surgery — Surgical procedure performed using an operating endoscope that is introduced into the body through a natural orifice and is then passed into the peritoneal cavity through the lumen of an organ such as the stomach, bowel or vagina.
  Other Names: Natural Orifice Transluminal Endoscopic Surgery
  Arms: Transvaginal Laparoscopic-Assisted Colectomy

SUMMARY:
This study aims to prospectively evaluate a laparoscopic-assisted transvaginal approach for colonic resection in adult women that eliminates the need for an abdominal incision to remove surgical specimens. It is hypothesized that this LANOS technique will improve patient outcomes such as postoperative surgical site infection (SSI) rates, thereby improving patient satisfaction and also reducing hospital length-of-stay and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥ 18 years of age
2. Diagnosed with one of the following benign or malignant conditions for which they require colonic resection with a specimen that may be removed transvaginally if randomized to that group:

   * Adenomatous polyposis
   * Chronic GI bleeding
   * Chronic obstruction
   * Colon cancer
   * Colonic inertia
   * Diverticular disease
   * Rectal cancer
   * Colorectal Polyps
   * Rectal prolapse
   * Slow transit constipation / colonic inertia
3. Require one of the following elective operations that may be safely performed by current laparoscopic-assisted techniques:

   * Right hemicolectomy
   * Left hemicolectomy
   * Subtotal colectomy
   * Total abdominal colectomy
   * Sigmoid colectomy
   * Rectosigmoid resection
   * Low anterior resection
4. Willingness and ability to comply with the requirements of the study protocol including follow-up
5. Willingness and ability to sign the study specific informed consent

Exclusion Criteria:

1. Current pregnancy or considering becoming pregnant during the follow-up period or within 6 months of surgery
2. Any anatomical consideration that in the Investigator's opinion would make the traditional laparoscopic or transvaginal approach to resection excessively risky or impossible. Patients with bulky tumors that would require open operations are not candidates for this study.
3. Body Mass Index (BMI) > 35
4. Vaginal stenosis
5. Prior reconstructive surgery of the vagina not including hysterectomy
6. ASA classes 4 and 5
7. Advanced renal insufficiency (estimated creatinine clearance ≤30 mL/min/1.73 m2)
8. Any history of pelvic radiation
9. Anticipated need for an ostomy at the time of operation
10. Patients requiring urgent or emergent surgery
11. Patients with prior or suspected diagnosis of inflammatory bowel disease such as Crohns disease or ulcerative colitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-operative Infections | Post-operative day 1 through 1 year
  To evaluate the effects of a laparoscopic-assisted transvaginal colonic resection on postoperative recovery, as measured primarily by surgical site infection rates, compared to standard laparoscopic-assisted colonic resection.

SECONDARY OUTCOMES:
Post-operative Pain | Post-operative day 1 through 1 year
  1. Pain score assessments: The investigator's staff will provide a rating scale to the patients to self-rate and record their pain at baseline (prior to surgery), at 24, 48, 72, 96, 120, 144 and 168 hours following the procedure end time (or discharge if earlier), and at 14 ± 7 days, 30 ± 7 days, 60 ± 14 days, and 12 months ± 14 days postoperatively using a 10 point visual analogue and pain faces scale where 0 is for no pain and 10 is for the worst pain imaginable. . These data will be recorded using the Pain Assessment Form. In addition, the amount of narcotic pain medication administered through postoperative day 7 (or discharge if earlier) will be recorded and analyzed as morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Sanchez, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States